CLINICAL TRIAL: NCT00607711
Title: A Phase I Study of Oral Palifosfamide Tris in Advanced, Refractory, Solid Tumors
Brief Title: Study of Oral Palifosfamide Tris in Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: IND was withdrawn
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Brian Schwartz, MD Chief Medical Officer, ZIOPHARM Oncology, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPC1001
Record Dates: First submitted 2008-01-24; First posted 2008-02-06 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2008-01

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: oral palifosfamide tris

INTERVENTIONS:
Drug: oral palifosfamide tris — Capsule(s) given daily for 15 days followed by a 6 day rest. This is a dose escalation arm.

SUMMARY:
The study of maximum tolerated dose and safety of oral palifosfamide tris capsules in advanced, refractory, solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histological or cytological confirmation of advanced cancer that is refractory to standard therapies for their condition.
2. Men and women of ≥18 years of age.
3. Life expectancy of at least 12 weeks.
4. Eastern Cooperative Oncology Group (ECOG) performance score ≤2 (see Appendix 4).
5. Eligible subjects MUST have at least one measurable lesion as defined by RECIST guidelines. If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology. Measurable lesions must NOT have been in a previously irradiated field or injected with biological agents.
6. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements, to be conducted ≤2 weeks prior to Baseline:

   * Creatinine < 1.5× upper limit of normal (ULN) OR a calculated creatinine clearance ≥70 cc/min
   * Total bilirubin ≤2×ULN
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN
   * Granulocytes in peripheral blood ≥2.0×109/L, hemoglobin ≥8.5 g/dL, and platelets ≥50,000/µL
7. Written informed consent in compliance with ZIOPHARM policies and the Human Investigation Review Committee (IEC/IRB) having jurisdiction over the site.
8. Men and women of childbearing potential must use effective contraception from Screening through his/her duration of study participation.
9. Women of childbearing potential must have a negative serum pregnancy test prior to entering the study.

Exclusion Criteria:

1. New York Heart Association (NYHA) functional Class ≥III myocardial infarction (see Appendix 5) within 6 months.
2. Uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation; a QTc ≥450 msec; or a ≥Grade 2 atrioventricular (AV) block or left bundle branch block (LBBB); or documented history of prolonged QTc.
3. Pregnancy and/or lactation.
4. Uncontrolled systemic infection (documented with microbiological studies).
5. Inadequate renal function as defined by the presence of one or more of the following:

   * Creatinine clearance (CrCl) <70 cc/min
   * Serum creatinine >1.5×ULN
   * Prior nephrectomy
   * Urinary tract obstruction
6. Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry (mitomycin C or nitrosureas should not be given within 6 weeks of study entry).
7. Radiotherapy during study or within 3 weeks of study entry.
8. Surgery within 4 weeks of start of study drug.
9. Other investigational drug therapy outside of this trial during or within 4 weeks of study entry.
10. History of invasive second primary malignancy diagnosed within the previous 3 years except for Stage I endometrial/cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer.
11. Substance abuse, medical, psychological, or social conditions that may interfere with the subject's participation in the study or evaluation of study results.
12. Any condition that is unstable or could jeopardize the safety of the subject and his/her compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Toxicities | 9 months

SECONDARY OUTCOMES:
Safety | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Shah, MD, Study Director — ZIOPHARM Oncology, Inc.